CLINICAL TRIAL: NCT05384041
Title: Cranial Electrotherapy Stimulation for the Treatment of Major Depressive Disorder in Adults
Acronym: CES-MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher Wallace Laboratories (Industry)
Collaborators: NAMSA (Other); Climb Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FW-200-05
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Depressive Disorder; Major Depressive Disorder; Cranial Electrotherapy Stimulation; FW-200
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Pivotal Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Remote, randomized, decentralized, controlled, triple-blind (subject, Principal Investigator, Sponsor) pivotal investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) (Active Comparator): The Fisher Wallace Stimulator provides cranial electrotherapy stimulation and is an active device.
  Interventions: Device: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device)
- Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device) (Placebo Comparator): The placebo device is designed to provide exactly the same patient experience as the active device; however, the placebo device will not deliver the same frequencies as the active device. The placebo device will provide no therapeutic benefit.
  Interventions: Device: Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)

INTERVENTIONS:
Device: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) — The indicated use in adults (ages 21-65 years) is for 20 minutes twice daily, upon waking for the day and at bedtime. The treatment period of the intervention will have a duration of four weeks.
  Other Names: Fisher Wallace Stimulator FW-200; FW-200
  Arms: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device)
Device: Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device) — The placebo device is designed to provide exactly the same patient experience as the active device; however, the placebo device will not deliver the same frequencies as the active device. The placebo device will provide no therapeutic benefit.
  Arms: Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)

SUMMARY:
This study is designed to evaluate the safety and efficacy of the Fisher Wallace Stimulator FW-200 to deliver Cranial Electrotherapy Stimulation (CES) for the treatment of moderate to severe Major Depressive Disorder (MDD) in adults.

DETAILED DESCRIPTION:
This prospective, fully remote, randomized, controlled, triple-blind (subject, Principal Investigator, Sponsor) pivotal study is designed to evaluate the safety and efficacy of the Fisher Wallace Stimulator FW-200 to deliver Cranial Electrotherapy Stimulation (CES) for the treatment of moderate to severe Major Depressive Disorder (MDD) in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years and a resident of the United States of America
2. Meets DSM-5 diagnostic criteria for moderate to severe Major Depressive Disorder
3. Baseline BDI-II score between 20 and 63, inclusive (in moderate to severe range)
4. Able to receive packages to their home via United Parcel Service/Fedex/United States Postal Service or other delivery service
5. Willing and able to send and receive study related text messages on an internet capable mobile device throughout the duration of the study
6. Owns and uses a personal, verifiable email address
7. Able to commit to two (2) 20-minute treatment sessions per day for 4 weeks, one treatment upon waking for the day and one treatment before going to bed
8. Willing to abstain from use of recreational drugs, hypnotics, steroids, and/or marijuana products through study completion
9. Willingness to not initiate treatment for a mental health issue during the course of the study
10. Fluent in English
11. Sexually active females of childbearing potential willing to commit to practicing at least one or more of the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception, or abstinence
12. In the opinion of the investigator, able to comply with study requirements and complete the study

Exclusion Criteria:

1. History of suicide attempt or active suicidal ideation with plan or intent in the past 30 days.
2. In the opinion of the investigator, considered high risk of suicide
3. Previous hospitalization or institutionalization for mental health condition within one year of study entry
4. Underwent electronic brain stimulation or neuromodulation within the past one year, including CES, transcranial magnetic stimulation, electroconvulsive therapy, and deep brain stimulation
5. Modification of prescription medications that affect the nervous system (e.g., psychotropic medications) within 30 days of study entry
6. Use of recreational drugs, hypnotics, steroids, and/or marijuana products in the past 30 days
7. History of alcohol use disorder or other substance use disorder in the past 12 months
8. Females currently pregnant or planning to conceive during study participation, or unwilling to comply with birth control requirements
9. Known history of heart disease
10. Known history of trigeminal neuralgia
11. Implanted with an electronic device such as a defibrillator, deep brain stimulator, or pacemaker
12. Unstable medical condition including any condition requiring hospitalization or change in treatment in the prior 30 days
13. Legally blind and/or deaf and without in-home care service to assist with study participation
14. Meets M.I.N.I. assessment criteria for, or has been diagnosed with, any of the following: Bipolar I disorder, bipolar II disorder, other specified bipolar and related disorder, panic disorder, agoraphobia, social anxiety disorder (social phobia), obsessive-compulsive disorder, posttraumatic stress disorder, alcohol use disorder in the past 12 months, substance use disorder (non-alcohol) in the past 12 months, any psychotic disorder (e.g., schizophrenia, schizoaffective disorder), major depressive disorder with psychotic features, anorexia nervosa, bulimia nervosa, binge-eating disorder, generalized anxiety disorder, any cognitive or developmental disorder (e.g., autism, Down's Syndrome), any personality disorder or psychiatric disorder that may interfere with study participation
15. Current participation in another investigational study or participated in an investigational study within the past 30 days
16. In the opinion of the investigator, may not be able to comply with study requirements
17. Any employee, family member, or personal associate of the Sponsor or their designees conducting the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Lapidus, MD, PhD, Principal Investigator
Locations (1):
- New York Neuromodulation Medical, PLLC, New York, New York, United States

REFERENCES:
- [Derived] Gehrman PR, Bartky EJ, Travers C, Lapidus K. A Fully Remote Randomized Trial of Transcranial Alternating Current Stimulation for the Acute Treatment of Major Depressive Disorder. J Clin Psychiatry. 2024 Apr 22;85(2):23m15078. doi: 10.4088/JCP.23m15078. PMID 38696220

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Started | 126 | 129
Completed | 121 | 125
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device) | Total
Number analyzed (Participants) | 126 | 129 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.04) | 40.1 (10.90) | 39.8 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 89 | 185
  Male | 30 | 40 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 92 | 99 | 191
  Asian | 4 | 5 | 9
  Black or African American | 9 | 7 | 16
  Hispanic or Latino | 9 | 7 | 16
  Other | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 126 | 129 | 255
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.5 (5.1) | 20.7 (5.6) | 20.6 (5.4)
Baseline Clinical Characteristics [Mean (Standard Deviation); unit: units on a scale]
  Beck Depression Inventory-II (BDI-II) | 34.1 (8.88) | 33.9 (8.99) | 34.0 (8.92)
  Personal Health Questionnaire Depression Scale (PHQ-9) | 16.0 (4.76) | 15.9 (4.82) | 16.0 (4.78)
  Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) | 16.0 (3.91) | 15.9 (3.67) | 16.0 (3.78)
Baseline Clinical Characteristics [Median (Full Range); unit: units on a scale]
  Beck Depression Inventory-II (BDI-II) | 33 [20 to 57] | 33 [20 to 59] | 33 [20 to 59]
  Personal Health Questionnaire Depression Scale (PHQ-9) | 16 [4 to 26] | 16 [6 to 27] | 16 [4 to 27]
  Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) | 16 [8 to 25] | 16 [8 to 25] | 16 [8 to 25]
Beck Depression Inventory-II (BDI-II) clinically based categories [Count of Participants; unit: Participants]
  Minimal (scores 0-13) | 0 | 0 | 0
  Mild (scores 14-19) | 0 | 0 | 0
  Moderate (scores 20-28) | 44 | 39 | 83
  Severe (scores 29-63) | 82 | 90 | 172
Use of concurrent anti-depressant medication [Count of Participants; unit: Participants] | 55 | 47 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change in the Beck Depression Inventory Second Edition (BDI-II) at Week Two Compared to Baseline.
Description: The Beck Depression Inventory Second Edition (BDI-II) is a multiple-choice self-report inventory that assesses severity of depression. The BDI-II contains 21 items on a 4-point scale from 0 (symptom absent) to 3 (severe symptoms). The minimum score is 0 and the maximum score is 63, with a higher score indicating more severe depressive symptoms.
  The candidate subject's BDI-II score must be within the range of 20 to 63 indicating moderate to severe Major Depressive Disorder.
Time Frame: Change at week two compared to baseline.
Population: Intent to Treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
units on a scale | 16.65 [14.691 to 18.610] | 14.36 [12.244 to 16.476]
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Intent to Treat analyses; Test type: Superiority; p = 0.056, Regression, Linear

2. Secondary Outcome: Change in the Beck Depression Inventory Second Edition (BDI-II) at Weeks One and Four Compared to Baseline.
Description: as for outcome 1
Time Frame: Change at weeks one and four compared to baseline.
Population: Intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
units on a scale
  Change in BDI-II at Week 1 (ITT analysis): number analyzed (Participants) | 124 | 125
  Change in BDI-II at Week 1 (ITT analysis) | 14.1 (9.93) | 11.5 (10.68)
  Change in BDI-II at Week 4 (ITT analysis): number analyzed (Participants) | 121 | 125
  Change in BDI-II at Week 4 (ITT analysis) | 19.9 (11.91) | 16.9 (12.46)
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active - Control) at Week 1; Test type: Superiority; p = 0.048, t-test, 2 sided

3. Secondary Outcome: Change in the Patient Health Questionnaire-9 (PHQ-9) at Weeks One, Two, and Four Compared to Baseline.
Description: The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale covering the Diagnostic and Statistical Manual, 5th Edition (DSM-5) for Major Depressive Disorder, with a diagnostic algorithm and score-based assessment of presence and severity of depression. The minimum score is 0 and the maximum score is 27, with a higher score indicating more severe depressive symptoms.
Time Frame: Change at weeks one, two, and four compared to baseline.
Population: Intent to Treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
units on a scale
  Change in PHQ-9 at Week 1 | 5.27 [4.338 to 6.211] | 4.50 [3.533 to 5.475]
  Change in PHQ-9 at Week 2 | 7.46 [6.457 to 8.470] | 6.29 [5.144 to 7.432]
  Change in PHQ-9 at Week 4 | 8.88 [7.823 to 9.946] | 7.72 [6.559 to 8.881]
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.2595, t-test, 2 sided
Statistical Analysis 2: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.1286, t-test, 2 sided
Statistical Analysis 3: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.1449, t-test, 2 sided

4. Secondary Outcome: Change in the Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR) at Weeks One, Two, and Four Compared to Baseline.
Description: The Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR) is a 16-item rating scale that assesses nine criterion symptom domains to diagnose a major depressive episode. The minimum score is 0 and the maximum score is 27, with a higher score indicating more severe depressive symptoms.
Time Frame: Change at weeks one, two, and four compared to baseline.
Population: Intent to Treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
units on a scale
  Change in QIDS-SR at Week 1 | 5.53 [4.688 to 6.377] | 4.77 [3.923 to 5.613]
  Change in QIDS-SR at Week 2 | 6.72 [5.842 to 7.589] | 5.71 [4.719 to 6.705]
  Change in QIDS-SR at Week 4 | 7.99 [7.038 to 8.946] | 6.90 [5.938 to 7.870]
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.2065, t-test, 2 sided
Statistical Analysis 2: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.1349, t-test, 2 sided
Statistical Analysis 3: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.1142, t-test, 2 sided

5. Secondary Outcome: Beck Depression Inventory Second Edition (BDI-II) Responder Rate by Time Point (% of Subjects With a 50% or Better Improvement in Score From Baseline).
Description: as for outcome 1
Time Frame: Four weeks following baseline.
Population: Intent-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
Participants
  Week 1 Response: Yes | 46 | 38
  Week 1 Response: No | 80 | 91
  Week 2 Response: Yes | 64 | 55
  Week 2 Response: No | 62 | 74
  Week 4 Response: Yes | 82 | 68
  Week 4 Response: No | 44 | 61
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.231, Chi-squared
Statistical Analysis 2: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.192, Chi-squared
Statistical Analysis 3: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.045, Chi-squared

6. Post Hoc Outcome: Change in the Beck Depression Inventory Second Edition (BDI-II) at Weeks One and Four Compared to Baseline (Per Protocol).
Description: as for outcome 1
Time Frame: Change at weeks one and four compared to baseline.
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 126 | 129
units on a scale
  Change in BDI-II at Week 1 (Per protocol analysis): number analyzed (Participants) | 117 | 117
  Change in BDI-II at Week 1 (Per protocol analysis) | 14.4 (10.14) | 11.3 (10.09)
  Change in BDI-II at Week 4 (Per protocol analysis): number analyzed (Participants) | 99 | 101
  Change in BDI-II at Week 4 (Per protocol analysis) | 20.0 (11.87) | 16.5 (12.47)

7. Post Hoc Outcome: Change in the Beck Depression Inventory Second Edition (BDI-II) at Week Two Compared to Baseline (Per Protocol).
Description: as for outcome 1
Time Frame: Change at week two compared to baseline.
Population: Per protocol (PP) population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
Number analyzed (Participants) | 109 | 108
units on a scale | 17.15 [15.040 to 19.253] | 13.62 [11.439 to 15.802]
Statistical Analysis 1: Comparison: Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) vs Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device); Test type: Superiority; p = 0.005, Regression, Linear

8. Post Hoc Outcome: Change in BDI-II From Baseline at Weeks 1, 2, and 4, Stratified by Gender (ITT Analysis)
Description: as for outcome 1
Time Frame: Change at weeks 1, 2, and 4 compared to baseline
Population: Intent to Treat population (N = 255)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Female (Active Device); Male (Active Device): The Fisher Wallace Stimulator provides cranial electrotherapy stimulation and is an active device.
- Female (Placebo Device); Male (Placebo Device): The placebo device is designed to provide exactly the same patient experience as the active device; however, the placebo device will not deliver the same frequencies as the active device. The placebo device will provide no therapeutic benefit.
- Total (Female): Total females across active and placebo arms
- Total (Males): Total males across active and placebo arms
Arm/Group | Female (Active Device) | Female (Placebo Device) | Total (Female) | Male (Active Device) | Male (Placebo Device) | Total (Males)
Number analyzed (Participants) | 95 | 85 | 180 | 29 | 40 | 69
units on a scale
  Week 1 | 15 [13.032 to 16.884] | 10.6 [8.485 to 12.692] | 12.9 [11.451 to 14.338] | 11.5 [7.265 to 15.701] | 13.6 [9.634 to 17.516] | 12.7 [9.865 to 15.526]
  Week 2: number analyzed (Participants) | 94 | 85 | 179 | 29 | 40 | 69
  Week 2 | 17.9 [15.844 to 19.986] | 14.2 [11.723 to 16.583] | 16.1 [14.534 to 17.723] | 12.6 [7.702 to 17.401] | 14.8 [10.503 to 19.097] | 13.9 [10.707 to 17.003]
  Week 4: number analyzed (Participants) | 92 | 85 | 177 | 29 | 40 | 69
  Week 4 | 21.2 [18.855 to 23.536] | 17.1 [14.515 to 19.603] | 19.2 [17.474 to 20.944] | 15.6 [10.648 to 20.524] | 16.5 [12.025 to 20.925] | 16.1 [12.873 to 19.330]
Statistical Analysis 1: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.0026, Regression, Linear
Statistical Analysis 2: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.4706, Regression, Linear
Statistical Analysis 3: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.0197, Regression, Linear
Statistical Analysis 4: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.4858, Regression, Linear
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.0183, Regression, Linear
Statistical Analysis 6: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.7885, Regression, Linear

9. Post Hoc Outcome: Change in BDI-II From Baseline at Weeks 1, 2, and 4, Stratified by Gender (Per Protocol Analysis)
Description: as for outcome 1
Time Frame: Change at weeks 1, 2, and 4 compared to baseline
Population: Per protocol population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Female (Active Device) | Female (Placebo Device) | Male (Active Device) | Male (Placebo Device)
Number analyzed (Participants) | 74 | 64 | 23 | 37
units on a scale
  Week 1 | -15.22 [-17.28 to -13.27] | -9.79 [-12.00 to -7.59] | -14.27 [-17.96 to -10.58] | -12.47 [-15.37 to -9.57]
  Week 2 | -18.23 [-20.49 to -15.97] | -13.76 [-16.18 to -11.33] | -15.53 [-19.60 to -11.47] | -13.49 [-16.69 to -10.30]
  Week 4 | -21.53 [-24.01 to -19.05] | -17.04 [-19.70 to -14.38] | -17.92 [-22.38 to -13.26] | -15.25 [-18.76 to -11.75]
Statistical Analysis 1: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p < 0.001, Regression, Linear
Statistical Analysis 2: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.450, Regression, Linear
Statistical Analysis 3: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.008, Regression, Linear
Statistical Analysis 4: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.438, Regression, Linear
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.016, Regression, Linear
Statistical Analysis 6: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.355, Regression, Linear

10. Post Hoc Outcome: Change in PHQ-9 From Baseline at Weeks 1, 2, and 4, Stratified by Gender (Per Protocol Analysis)
Description: as for outcome 3
Time Frame: Change at weeks 1, 2, and 4 compared to baseline
Population: Per protocol population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Female (Active Device) | Female (Placebo Device) | Male (Active Device) | Male (Placebo Device)
Number analyzed (Participants) | 74 | 64 | 23 | 37
units on a scale
  Week 1 | -5.42 [-6.49 to -4.35] | -3.82 [-4.97 to -2.67] | -6.13 [-8.05 to -4.21] | -4.97 [-6.48 to -3.45]
  Week 2 | -7.84 [-9.02 to -6.65] | -6.12 [-7.39 to -4.85] | -8.00 [-10.13 to -5.87] | -5.85 [-7.53 to -4.17]
  Week 4 | -9.48 [-10.61 to -8.35] | -8.32 [-9.53 to -7.11] | -8.80 [-10.82 to -6.77] | -6.77 [-8.36 to -5.18]
Statistical Analysis 1: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.046, Regression, Linear
Statistical Analysis 2: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.351, Regression, Linear
Statistical Analysis 3: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.053, Regression, Linear
Statistical Analysis 4: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.120, Regression, Linear
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.170, Regression, Linear
Statistical Analysis 6: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.122, Regression, Linear

11. Post Hoc Outcome: Change in QIDS From Baseline at Weeks 1, 2, and 4, Stratified by Gender (Per Protocol Analysis)
Description: as for outcome 4
Time Frame: Change at weeks 1, 2, and 4 compared to baseline
Population: Per protocol population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Female (Active Device) | Female (Placebo Device) | Male (Active Device) | Male (Placebo Device)
Number analyzed (Participants) | 74 | 64 | 23 | 37
units on a scale
  Week 1 | -5.79 [-6.76 to -4.82] | -4.33 [-5.37 to -3.29] | -5.91 [-7.65 to -4.16] | -5.55 [-6.92 to -4.18]
  Week 2 | -7.46 [-8.49 to -6.42] | -5.52 [-6.64 to -4.41] | -6.52 [-8.38 to -4.65] | -5.31 [-6.78 to -3.85]
  Week 4 | -8.53 [-9.59 to -7.46] | -7.45 [-8.59 to -6.30] | -8.21 [-10.12 to -6.30] | -6.40 [-7.90 to -4.90]
Statistical Analysis 1: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.044, Regression, Linear
Statistical Analysis 2: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.751, Regression, Linear
Statistical Analysis 3: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.013, Regression, Linear
Statistical Analysis 4: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.318, Regression, Linear
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.173, Regression, Linear
Statistical Analysis 6: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.142, Regression, Linear

12. Post Hoc Outcome: Subgroup Analysis - Proportion of Subjects Achieving at Least 50% Improvement From Baseline in BDI-II (ITT Analyses)
Description: as for outcome 1
Time Frame: Weeks 1, 2, and 4 following baseline
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Female (Active Device) | Female (Placebo Device) | Male (Active Device) | Male (Placebo Device)
Number analyzed (Participants) | 95 | 85 | 29 | 40
Participants
  Week 1 | 37 | 20 | 9 | 18
  Week 2: number analyzed (Participants) | 94 | 85 | 29 | 40
  Week 2 | 52 | 35 | 12 | 20
  Week 4: number analyzed (Participants) | 92 | 85 | 29 | 40
  Week 4 | 68 | 47 | 14 | 21
Statistical Analysis 1: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.026, Chi-squared
Statistical Analysis 2: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.241, Chi-squared
Statistical Analysis 3: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.059, Chi-squared
Statistical Analysis 4: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.478, Chi-squared
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.009, Chi-squared
Statistical Analysis 6: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.729, Chi-squared

13. Post Hoc Outcome: Subgroup Analysis - Proportion of Subjects Achieving at Least 50% Improvement From Baseline in BDI-II (Per Protocol Analyses)
Description: as for outcome 1
Time Frame: Weeks 1, 2, and 4 following baseline
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Groups:
- Total (Active Device): The Fisher Wallace Stimulator provides cranial electrotherapy stimulation and is an active device.
- Total (Placebo Device): The placebo device is designed to provide exactly the same patient experience as the active device; however, the placebo device will not deliver the same frequencies as the active device. The placebo device will provide no therapeutic benefit.
Arm/Group | Female (Active Device) | Female (Placebo Device) | Male (Active Device) | Male (Placebo Device) | Total (Active Device) | Total (Placebo Device)
Number analyzed (Participants) | 74 | 64 | 23 | 37 | 97 | 101
Participants
  Week 1 | 30 | 12 | 9 | 15 | 39 | 27
  Week 2 | 41 | 24 | 11 | 17 | 52 | 41
  Week 4 | 56 | 36 | 12 | 18 | 68 | 54
Statistical Analysis 1: Comparison: Total (Active Device) vs Total (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.044, Chi-squared
Statistical Analysis 2: Comparison: Total (Active Device) vs Total (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.067, Chi-squared
Statistical Analysis 3: Comparison: Total (Active Device) vs Total (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.016, Chi-squared
Statistical Analysis 4: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.006, Chi-squared
Statistical Analysis 5: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.036, Chi-squared
Statistical Analysis 6: Comparison: Female (Active Device) vs Female (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.016, Chi-squared
Statistical Analysis 7: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 1; Test type: Superiority; p = 0.914, Chi-squared
Statistical Analysis 8: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 2; Test type: Superiority; p = 0.887, Chi-squared
Statistical Analysis 9: Comparison: Male (Active Device) vs Male (Placebo Device); Difference (Active-Control) at Week 4; Test type: Superiority; p = 0.791, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning through the end of the treatment period for a total of four weeks per trial participant.
Description: On each day of trial therapy through study completion, participants reported in ePRO whether or not they used the study device as instructed and if there had been a change to their health status or medications over the previous 24 hours. A free text form allowed participants to describe any changes to their health, including any adverse events, during trial therapy.
Arm/Group | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/129
Other Adverse Events (participants affected / at risk) | 19/126 | 10/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fisher Wallace Cranial Electrotherapy Stimulator (Active Device) (N=126) | Fisher Wallace Cranial Electrotherapy Stimulator (Placebo Device) (N=129)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Headache / Anxiety (General disorders) | 1 | 0
Headache / Allergy (General disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 3
Decreased appetite (Gastrointestinal disorders) | 1 | 1
Vision blurred / Allergy (General disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinusitis (Infections and infestations) | 2 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Photopsia (Eye disorders) | 1 | 0
Photopsia / Skin discomfort (General disorders) | 1 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Eye movement disorder / Skin discomfort (General disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 3 | 0
Poor quality sleep (Nervous system disorders) | 2 | 2
Abnormal dreams (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT05384041/Prot_SAP_000.pdf